CLINICAL TRIAL: NCT06179043
Title: Examining the Impact of Different Types of Front-of-package Warning Labels for Sugar-sweetened Beverages on Perceived Weight Stigmatization Among a Sample of US Adults
Brief Title: Impact of Front-of-package Warning Labels on Perceived Weight Stigmatization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 23-3069
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Weight Stigma
MeSH Terms: conditions — Weight Prejudice

STUDY DESIGN:
Intervention Model Description: Between-subjects intervention: label type (4 arms); Within-subjects intervention: regular or weight-neutral version of label (2 versions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control labels (Sham Comparator): Individuals in this trial arm will see neutral control labels on sugar-sweetened beverages.
  Interventions: Behavioral: Control labels
- Nutrient warning labels (Experimental): Individuals in this trial arm will see nutrient warning labels on sugar-sweetened beverages.
  Interventions: Behavioral: Nutrient warning labels
- Text-only health warning labels (Experimental): Individuals in this trial arm will see text-only health warning labels on sugar-sweetened beverages.
  Interventions: Behavioral: Text-only health warning labels
- Graphic warning labels (Experimental): Individuals in this trial arm will see graphic health warning labels on sugar-sweetened beverages.
  Interventions: Behavioral: Graphic health warning labels

INTERVENTIONS:
Behavioral: Nutrient warning labels — In random order, participants in this arm will see an image of fictional sugar-sweetened beverages carrying:
  * Labels that read "high in sugars" and "high in calories"
  * A label that reads "high in sugars"
  Arms: Nutrient warning labels
Behavioral: Text-only health warning labels — In random order, participants in this arm will see an image of fictional sugar-sweetened beverages carrying:
  * A label that reads "Drinking beverages with added sugars contributes to obesity, type 2 diabetes and tooth decay"
  * A label that reads "Drinking beverages with added sugars contributes type 2 diabetes and tooth decay"
  Arms: Text-only health warning labels
Behavioral: Graphic health warning labels — In random order, participants in this arm will see an image of fictional sugar-sweetened beverages carrying:
  * A label that reads "Drinking beverages with added sugars contributes to obesity, type 2 diabetes and tooth decay" and contains graphics illustrating obesity, type 2 diabetes, and tooth decay
  * A label that reads "Drinking beverages with added sugars contributes type 2 diabetes and tooth decay" and contains graphics illustrating type 2 diabetes and tooth decay
  Arms: Graphic warning labels
Behavioral: Control labels — In random order, participants in this arm will see an image of fictional sugar-sweetened beverages carrying:
  * A neutral bar code label
  * A neutral quick response (QR) code label (not scannable)
  Arms: Control labels

SUMMARY:
The goal of this experiment is to examine the effects of three different types of front-of-package warning labels for sugar-sweetened beverages on perceived weight stigmatization, as well as the effect of making such labels more weight-neutral. The main questions this experiment aims to answer are:

* Are certain types of front-of-package warning labels perceived as more stigmatizing than others?
* Are more weight-neutral versions of front-of-package warning labels perceived as less stigmatizing than their regular versions?
* Is there a trade-off between label effectiveness in discouraging product consumption and perceived weight stigmatization?

Additionally, this experiment also aims to answer the following questions:

* Does exposure to certain types of front-of-package warning labels lead to changes in participants' weight bias?
* Are changes in participants' weight bias as a result of label exposure mediated by attribution of personal responsibility for body weight, pathogen disgust, or perceived social consensus?

DETAILED DESCRIPTION:
Participants will be randomly assigned to see one of four types of labels: control labels, nutrient warning labels, text-only health warning labels, or graphic health warning labels. Participants will then see an image depicting different types of fictional sugar-sweetened beverages carrying the label type that they were assigned to. Participants will see this image twice, in random order, each time differing in whether the label is weight-neutral or not (i.e., whether the label references calories/obesity or not). Each time, participants will answer survey questions about the label. Last, participants will answer survey questions measuring their weight bias and potential mediating variables.

ELIGIBILITY:
Inclusion criteria:

* At least 21 years of age.
* Residing in the US.

Exclusion Criteria:

-Involved in any pre-testing.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2522 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Perceived weight stigmatization, mean score | Immediately after exposure to intervention (i.e., study stimuli), assessed during one-time online study survey.
  Stigmatization of people with obesity will be measured by survey through a three-item scale. Items will inquire about how much participants perceive the label to (1) stigmatize people with obesity, (2) promote negative stereotypes about people with obesity, and (3) portray people with obesity in a disrespectful manner. Response options will be on a 1 to 5 scale, with higher scores representing a higher perceived weight stigmatization by the study labels. Each participant's responses to each item will be combined to obtain their final score on the outcome.

SECONDARY OUTCOMES:
Perceived message effectiveness, mean score | Immediately after exposure to intervention (i.e., study stimuli), assessed during one-time online study survey.
  How much the labels discourage participants from wanting to consume the products will be measured by survey. Response options will be on a 1 to 5 scale, with higher scores representing a higher perceived message effectiveness.
Weight bias, mean score | Immediately after exposure to intervention (i.e., study stimuli), assessed during one-time online study survey.
  Weight bias will be measured by survey through a seven-item scale. Items will present participants with adjective pairs and ask that they select the box closest to the adjective that they feel best describe their feelings and beliefs about people with obesity: (1) lazy-industrious, (2) no will power - has will power, (3) good self-control - poor self-control, (4) active - inactive, (5) self-indulgent - self-sacrificing, (6) dislikes food - likes food, (7) undereats - overeats. Response options will be 5 boxes between adjectives, which will be coded on a 1 to 5 scale so that higher scores represent higher weight bias. Each participant's responses to each item will be combined to obtain their final score on the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Aline D'Angelo Campos, MPP, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset and analytic code will be uploaded to a public repository upon publication of the study.
Supporting Information: Analytic Code
Time Frame: Upon publication of the study.
Access Criteria: No access criteria. The dataset and analytic code will be made publicly available at Open Science Framework.

REFERENCES:
- [Background] Grummon AH, Gibson LA, Musicus AA, Stephens-Shields AJ, Hua SV, Roberto CA. Effects of 4 Interpretive Front-of-Package Labeling Systems on Hypothetical Beverage and Snack Selections: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2333515. doi: 10.1001/jamanetworkopen.2023.33515. PMID 37703015
- [Background] Hayward LE, Vartanian LR. Potential unintended consequences of graphic warning labels on sugary drinks: do they promote obesity stigma? Obes Sci Pract. 2019 Aug 2;5(4):333-341. doi: 10.1002/osp4.353. eCollection 2019 Aug. PMID 31452918
- [Derived] D'Angelo Campos A, Grummon AH, Ng SW, Puhl RM, Golden SD, Hall MG. Front-of-Package Food Labels and Perceived Weight Stigmatization: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2516821. doi: 10.1001/jamanetworkopen.2025.16821. PMID 40540266

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT06179043/Prot_SAP_000.pdf